CLINICAL TRIAL: NCT06957535
Title: Community-led Navigation to Address Disparities in Mammography Among Native American Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Genentech Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00031873
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEAM (Active Comparator): TEAM (Tablet-based Education to improve the Acceptance of Mammography)
  Interventions: Behavioral: TEAM
- TEAM + Navigation (Experimental): TEAM (Tablet-based Education to improve the Acceptance of Mammography) and Navigation (provision of 1:1 support from a Diné peer-navigator)
  Interventions: Behavioral: Navigation; Behavioral: TEAM

INTERVENTIONS:
Behavioral: Navigation — Navigation is provision of 1:1 support from a Diné peer-navigator
  Arms: TEAM + Navigation
Behavioral: TEAM — TEAM encompasses culturally tailored mammography education modules

SUMMARY:
The goal of this study is to evaluate the effectiveness of an intervention to promote breast cancer screening mammography among women in one community on the Navajo Nation. The intervention is Tablet-based Education to improve the Acceptance of Mammography (TEAM). TEAM encompasses culturally-tailored mammography education modules that were developed using a community-based participatory research process. Women will be randomized to receive TEAM or TEAM + Navigation. Navigation involves monthly 1:1 support from a Diné peer-navigator.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as American Indian or Alaska Native (AIAN)
* Identify as Female
* Are 40-74 years of age
* Are a registered patient at Chinle Comprehensive HealthCare Facility (CCHFC)
* Live within 80 miles of CCHFC
* Have not received a mammogram within the prior 12 months
* Do not have a personal history of breast cancer
* Are not planning to move in the next 6 months
* Willing to be randomized

Exclusion Criteria:

* Do not self-identify as American Indian or Alaska Native (AIAN)
* Do not identify as Female
* Are not 40-74 years of age
* Are not a registered patient at CCHCF
* Do not live within 80 miles of CCHCF
* Have received a mammogram within the prior 12 months
* Have a personal history of breast cancer
* Are planning to move in the next 6 months
* Unwilling to be randomized

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as female
Enrollment: 200 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with mammography | 3 months post baseline
  Mammography uptake within 3 months of referral

CONTACTS AND LOCATIONS:
Overall Officials: Katie Nelson, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Navajo Nation Center for Indigenous Health, Chinle, Arizona, United States

IPD SHARING:
Plan to Share IPD: No